CLINICAL TRIAL: NCT02785718
Title: The Influence of the Proteins of the Contact Activation System on Thrombus Formation in Human Blood
Brief Title: The Proteins of the Contact Activation System
Acronym: CONTACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012.785
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Factor XI Deficiency; Factor XII Deficiency
Keywords: Contact system; Factor XI deficiency; Factor XII deficiency; Global haemostasis assays
MeSH Terms: conditions — Factor XI Deficiency; Factor XII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with FXI or FXII deficiency (Experimental): 12 patients with FXI deficiency and 6 patients with FXII deficiency
  Interventions: Other: Global Haemostasis assays

INTERVENTIONS:
Other: Global Haemostasis assays

SUMMARY:
Cardiovascular diseases are important causes of morbidity and mortality in the industrialized world. Abnormalities in the coagulation system, causing a hypercoagulable state, are a known risk factor for arterial and venous thrombosis. The contact activation system is part of the coagulation system and consists of four proteins: coagulation factor XII (FXII), FXI, prekallikrein and high molecular weight kininogen (HMWK). Clinical studies indicate an important role for the contact activation system on the risk of arterial thrombosis. Furthermore, there is substantial evidence from mouse studies that FXII and FXI participate in the formation and stability of thrombi. In vitro studies show that collagen, present in the vascular wall, is able to activate FXII and hereby stimulate thrombin formation and potentiate the formation of platelet-fibrin thrombi and FXIIa is able to change the structure of fibrin clots by binding to fibrin(ogen) and by generation of additional thrombin. However, the contact system also participates in the process of fibrinolysis, which degrades thrombi.

The investigators would like to investigate the contribution of the contact activation system to the formation of thrombi. The formation of a thrombus within the vascular bed is the main cause for occlusion of an artery or vein, which can lead to an infarct such as a heart attack. Due to the other functions of the contact system it is important to fully understand how the contact system contributes to thrombus formation, before it can be used as a target in the treatment of arterial thrombosis. The aim of this study is to determine the contribution of the proteins of the contact system, mainly FXII and FXI, in the platelet mediated formation and degradation of thrombi. This will be studied in flow models (perfusion-flow model and Chandler loop), in a static model (ROTEM®) and using thrombin generation assay.

ELIGIBILITY:
Inclusion Criteria:

* Deficiency in coagulation factor XII and factor XI (factor level<5%)
* Subjects of both gender
* Age ≥18 and ≤ 65
* Written informed consent from the subject
* Subject with a social security plan or beneficiary of such a plan.

Exclusion Criteria:

* Age below 18
* Age above 65
* Other known abnormalities of the coagulation system
* Thrombocytopenia
* Known platelet disorders
* Personal history of severe liver diseases
* Symptoms of active disease (e.g. cancer)
* The use of antiplatelet drugs
* The use of drugs that interfere with coagulation
* Ongoing diagnosed pregnancy upper 3 months
* Adult patients protected by law
* Concomitant participation to a biomedical research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
fibrinolytic degradation rate of the formed clots by ROTEM analysis | 1 day (cross sectional)

SECONDARY OUTCOMES:
the ex-vivo formation of platelet-mediated thrombi on collagen in a perfusion flow mode | 1 day (cross sectional)
biochemical composition of the thrombi formed in the Chandler loop | 1 day (cross sectional)
endogenous thrombin potential (ETP) of the platelet rich plasma of these patients | 1 day (cross sectional)

CONTACTS AND LOCATIONS:
Locations (1):
- Unité d'Hémostase Clinique Hôpital Louis Pradel, Bron, France